CLINICAL TRIAL: NCT06148103
Title: Sedation for Colonoscopy Procedures Using Dexmedetomidine Versus Propofol-Fentanyl Infusions: A Prospective Randomized Controlled Trial
Brief Title: A Comparison Between Dexmedetomidine and Propofol-fentanyl Infusions for Sedation for Colonoscopy Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zulekha Hospitals (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00385
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D group (Other): Patients who received Dexmedetomidine. The starting dose of dexmedetomidine was 1 microgram/kg over a period of 10 minutes, and then a maintenance infusion was titrated in a range from 0.2-1 μg/kg/h).
  Interventions: Drug: Patients who received Dexmedetomodine
- PF group (Other): Patients who received Propofol-Fentanyl infusions. Continued infusions of both fentanyl and propofol were 0.01-0.05 μg kg/ min 25-150 mg/h respectively.
  Interventions: Drug: patients who received propofol-fentanyl

INTERVENTIONS:
Drug: Patients who received Dexmedetomodine — 1 microgram/kg over a period of 10 minutes, and then a maintenance infusion was titrated in a range from 0.2-1 μg/kg/h).
  Other Names: D group
  Arms: D group
Drug: patients who received propofol-fentanyl — Continued infusions of both fentanyl and propofol were 0.01-0.05 μg kg/ min 25-150 mg/h respectively.
  Other Names: PF group
  Arms: PF group

SUMMARY:
Background: Different intravenous sedative drugs have been utilized for colonoscopy, with many anesthetists for painless sedation or monitored anesthesia care. The aim of this study was the quality of colonoscopy and the incidence of adverse events such as respiratory depression, hemodynamic instability, and failure to provide adequate sedation.

DETAILED DESCRIPTION:
Background: Different intravenous sedative drugs have been utilized for colonoscopy, with many anesthetists for conscious sedation or monitored anesthesia care. Aim of this study was the quality of colonoscopy and the incidence of adverse events such as respiratory depression, hemodynamic instability, and failure to provide adequate sedation.

Patients and methods: Sixty patients of both sexes and 21-60 years old with ASA physical status I-II, were randomly assigned to receive either dexmedetomidine (D group) or propofol-fentanyl (PF group) infusions in equal numbers. Minimal infusion rates of dexmedetomidine (0.1-0.4 μg/kg/h) in the D group and fentanyl (0.01-0.05 μg/kg/min) in the PF group were continued during colonoscopy, which lasted approximately 30 minutes.

ELIGIBILITY:
* Inclusion Criteria:

  1. both sexes
  2. 21-60 years old, with
  3. ASA physical status -
* Exclusion Criteria:

  * severe cardiovascular or respiratory disease
  * (ASA grade ≥III)
  * pregnancy
  * allergies to the drugs being used
  * known alcohol or substance abuse
  * expected communication difficulties with the patient.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
The quality of painless sedation during colonoscopy. | From start of procedure to 120 minutes after end of colonoscopy
  The patient's ability to cooperate and perform the procedure was evaluated using a 10-point numerical rating scale (NRS).

SECONDARY OUTCOMES:
incidence of adverse events, Prevalence of adverse effects | from start of procedure to 120 minutes after end of colonoscopy
  incidence of adverse events, hemodynamic instability, failure to provide adequate sedation.

CONTACTS AND LOCATIONS:
Overall Officials: sameh H Seyam, professor, Principal Investigator — Assistant professor, Anesthesiology, Intensive care and pain management
Locations (1):
- Al-Azhar faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No